CLINICAL TRIAL: NCT06027138
Title: Comparative Effects of Blood Flow Resistance and Slow Motion Strength Training on Explosive Power and Lower Limb Function Among Wrestlers.
Brief Title: Comparison Between Blood Flow Resistance and Slow Motion Strength Training in Wrestlers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC\RCR&AHS\23\0416
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Sports
Keywords: Strength training, BFR training, explosive power

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- blood flow resistance training (Active Comparator): vertical jump test
  1RM tests times pull ups and push ups test
  Interventions: Other: blood flow resistance training; Other: slow motion strength training
- slow motion strength training (Experimental): vertical jump test
  1RM tests times pull ups and push ups test
  Interventions: Other: blood flow resistance training; Other: slow motion strength training

INTERVENTIONS:
Other: blood flow resistance training — Muscle size and explosive power was determined by measuring the diameter of its arm and thigh muscles and performing 1RM testing in barbell parallel back squats and foot barbell Bench press ,vertical jump test and timed push ups and pull up tests .secondly treat the arm and thigh muscles to to blood flow resistance training and is administered for approx 2 months a frequency of four times per week at an intensity of seventy five to eight five percent for 4 to 12 reps,1 to 5 sets, at interval of 30 to 40 sec.then determine the impact of treatmnt measurement was again carried out on the circumference and explosive strength of arm and thigh muscles.
Other: slow motion strength training — We will use slow motion strength training method. Each exercise is performed by lifting weights for approximately 10 seconds, lowering the weight for another 10 seconds, and not resting between repetitions.before receiving treatment sample muscle size and explosive strength was determined by measuring the diameter of its arm and thigh muscles and performing 1RM testing in barbell parallel back squats and foot barbell Bench press (pre test).secondly treat the arm and thigh muscles to to slow motion weight training.weight training and is administered for approx 2 months a frequency of four times per week at an intensity of seventy five to eight five percent for 4 to 12 reps,1 to 5 sets, at interval of 30 to 40 sec.then determine the impact of treatmnt measurement was again carried out on the circumference and explosive strength of arm and thigh muscles. (Post test).

SUMMARY:
The sport of wrestling poses several challenges for strength and conditioning addressed by designing a resistance training program to meet these requirements. This Study provides recommendations for implementing an effective resistance training program for wrestlers.Blood Flow Restriction (BFR) training is a technique that combines low intensity exercise with blood flow occlusion that produces similar results to high intensity training. High-intensity, slow-motion strength training helps build muscle mass faster than lifting regular weights. This is because the slow-motion forces your muscles to hold the weight longer. With standard weightlifting, the faster the momentum, the less time your muscles are engaged.

This study will be conducted to compare effect of blood flow resistance and slow motion strength training on power and lower limb function among wrestler players.All subjects will be selected between age 18 to 35 years.Data will be collected from players in Pakistan sports board . Study design will be Randomized clinical trial. Measuring tape,1RM tests,vertical jump test and Timed push ups and pull ups test will be used to asses the power and lower limb function. Informed consent will be taken from All the participants.Athletes will be allocated randomly into two main groups.Group A and group B. On group A blood flow resistance training method will be performed and group B will be provided by slow motion strength training method to compare the effects of both techniques. Study will be conducted in nine months time period after the approval of synopsis. Data will be collected at the start of the research and after one year post research data will collected for analysis. SPSS will be used for data entry and analysis.

DETAILED DESCRIPTION:
Wrestling players will be allocated randomly into two main groups.On group A blood flow resistance training will be performed and Group B will be provided by slow motion strength training to compare the effects of both techniques During 1st visit of the patient these steps will be taken. A consent will be taken from athletes A complete thorough assessment will be done by researcher. The athletes will complete 1RM tests , vertical jump test ,Timed push-ups and pull ups test.

Techniques will then continue to selected subject according to their allocation In next visit. Patient will be reassessed by researcher. Sessions of techniques per week will be given.

Post training readings will be taken at the end of 6th week,total training will be of 6 weeks .

ELIGIBILITY:
Inclusion Criteria:

* Age:18 to 35 years
* Athletes registered at fitness center
* Athletes undergoing strength training program
* No history of previous ankle,knee,hip or back musculoskeletal condition that could influence their ability to perform 1RMtests and vertical jump tests

Exclusion Criteria:

* Athletes who will not have any systematic disease which can hinder the training.
* Athletes who would not commit to full participation in the study's training regime.
* Athletes have who have received surgery prior to study or undergone rehabilitation within the past year

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2023-03-25 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-08-22 (Estimated)

PRIMARY OUTCOMES:
measuring tape | 6 weeks
  Measurement of muscle size is often used to estimate muscle strength.For this purpose measuring tape is used to asses the skin fold thickness /muscle size
vertical jump test | 6 weeks
  The vertical jump test is a test of lower body power the athlete stands side on to a wall and reaches up with the hand closest to the wall. Keeping the feet flat on the ground, the point of the fingertips is marked or recorded. The athlete then stands away from the wall, and leaps vertically as high as possible using both arms and legs to assist in projecting the body upwards. The jumping technique can or cannot use a counter-movement. Attempt to touch the wall at the highest point of the jump. The difference in distance between the standing reach height and the jump height is the score. The best of three attempts is recorded
1RM tests | 6 weeks
  1. RM TESTS: The one repitition maximum is often considered as the gold standard for assessing the strength capacity of individuals in non laboratory environment.it is simply defined as maximum weight an individual can lift for only one repetition with correct technique
timed push ups and pull ups tests | 6 weeks
  The push-up fitness test (also called the press-up test) measures upper body strength and endurance. standard push-up begins with the hands and toes touching the floor, the body and legs in a straight line, feet slightly apart, the arms at shoulder-width apart, extended and at a right angle to the body. Keeping the back and knees straight, the subject lowers the body to a predetermined point, to touch the ground or some other object, or until there is a 90-degree angle at the elbows, then returns back to the starting position with the arms extended. This action is repeated without rest, and the test continues until exhaustion, or until they can do no more in rhythm or have reached the target number of push-ups Record the number of correctly completed push-ups

CONTACTS AND LOCATIONS:
Overall Officials: muzna munir, phd, Principal Investigator — Riphah International University
Locations (1):
- Pakistan sports board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No